CLINICAL TRIAL: NCT04108741
Title: Augmented Reality Treadmill Training in Patients With Parkinson's Disease: a Randomized Controlled Study
Brief Title: Augmented Reality Treadmill Training in Patients With Parkinson's Disease
Acronym: Falls_in_PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Veit Mylius, Priniciple Investigator, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V1 19.09.2019
Record Dates: First submitted 2019-09-20; First posted 2019-09-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Fall
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treadmill training with augmented reality dual tasking (Experimental)
  Interventions: Device: C-Mill augmented reality treadmill training
- treadmill training with random number generation dual tasking (Experimental)
  Interventions: Device: C-Mill augmented reality treadmill training
- treadmill training (Active Comparator)
  Interventions: Device: C-Mill augmented reality treadmill training

INTERVENTIONS:
Device: C-Mill augmented reality treadmill training — PD Patients will be randomized to treadmill training with augmented reality or to treadmill training with random number generation or to treadmill training for 3 weeks at 5 days a week for 30 minutes.

SUMMARY:
Gait disorder is a disabling symptom in Parkinson's disease (PD) affecting all patients during the course. Three methods of treadmill training (TT) will be compared to assess additional augmented reality (AR), or additional dual task (DT). AR TT, DT TT, and TT alone applied over 3 weeks at each day will be compared for their impact on falls, walking, freezing and attention for 3 months in a double blinded randomized controlled trial during regular neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Parkinson´s disease without dementia and hallucination
* at least one fall within the past 3 months or postural instability
* Gait disorder
* Hoehn and Yahr stages II-IV
* able to perform the treadmill therapy during a study

Exclusion Criteria:

* Contraindications to treadmill therapy (e.g. hip fracture)
* Dementia as defined by an Montreal cognitive assessment (MOCA) < 20

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of falls | 3 months before study to 3 months following the study
  group difference of the difference in falls

SECONDARY OUTCOMES:
Secondary outcomes: | before and after the training period of 3 weeks
  Freezing of Gait (FOG) Questionnaire
Sensor based gait analyses | before and after the training period of 3 weeks and after 3 months
  for one week

CONTACTS AND LOCATIONS:
Overall Officials: Veit Mylius, Prof. Dr., Principal Investigator — Department of Neurology, Kliniken Valens
Locations (1):
- Department of Neurology, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No